CLINICAL TRIAL: NCT01602419
Title: Surveillance of Safety and Efficacy of Wilate in Patients With Von Willebrand Disease
Status: Completed | Type: Observational
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: Wil-20
Record Dates: First submitted 2012-05-15; First posted 2012-05-21 (Estimated); Results first posted 2019-12-10 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients using Wilate as standard of care treatment: This patient population is being treated with Wilate as standard of care treatment
  Interventions: Other: Patients using Wilate as standard of care

INTERVENTIONS:
Other: Patients using Wilate as standard of care — Patients with von Willebrand Disease using Wilate for a period of 2 years.

SUMMARY:
This is an observational study, hence there is no study hypothesis

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of von Willebrand Disease who have been prescribed Wilate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: VWD patients of any gender, age, or VWD type
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (4):
  - Los Angeles Biomedical Research Institute, Torrance, California
  - Nicklaus Children's Hospital, Miami, Florida
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
- Fundación de la Hemofilia de Salta, Salta, Argentina
- Canada (9):
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. John Regional Hospital, Saint John, New Brunswick
  - Eastern Regional Health Authority, St. John's, Newfoundland and Labrador
  - McMaster University, Hamilton, Ontario
  - Queens University, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
- University Hospital Ostrava, Ostrava-Poruba, Czechia
- Werlhof-Institut, Hanover, Germany
- Centro Hospitalar Cova da Beira, Covilha, Portugal
- Spain (3):
  - Hospital Universitario de Burgos, Burgos
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Fundacion Jiminez Diaz, Madrid
- Skåne University Hospital, Malmo, Sweden
- Great Ormond Street Hospital for Children, London, United Kingdom
- Uruguay (2):
  - Hospital Pereira Rossell, Montevideo
  - Sanatorio Americano, Montevideo

RESULTS

PARTICIPANT FLOW:
Groups:
- Wilate: A total of 120 patients were enrolled in this study.
  Of the 120 patients enrolled into the study, 9 were excluded because they had not received any treatment with Wilate, leaving 111 patients in the safety (SAF) population. Of these 111 patients, 7 did not have a confirmed diagnosis of von Willebrand Disease (VWD) and 2 had another bleeding disorder, leaving 102 patients in the intention-to-treat (ITT) population. Of these 102 patients, 11 were excluded from the efficacy (EFF) population for the reasons summarised below.
Period: Overall Study
Arm/Group | Wilate
Started | 120
SAF Population | 111
ITT Population | 102
EFF Population | 91
Completed | 91
Not Completed | 29
Not completed — Not treated with Wilate | 9
Not completed — Adverse Drug Reaction | 4
Not completed — Insurance issues | 3
Not completed — Changed treatment centre | 1
Not completed — Treatment centre closed | 1
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Population: The SAF population consisted of 111 patients who received at least one dose of Wilate during the study.
Groups:
- SAF Population: Of the 120 patients enrolled in this study, 111 received at least one dose of Wilate and were included in the SAF population
Arm/Group | SAF Population
Number analyzed (Participants) | 111
Age, Continuous [Median (Full Range); unit: years]
  Age at study entry | 27 [0.8 to 83.2]
  Age at diagnosis of VWD | 13.5 [0 to 71.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 76
  Sex: Male | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic origin: Caucasian | 89
  Ethnic origin: Other | 17
  Ethnic origin: Asian | 3
  Ethnic origin: Black | 1
  Ethnic origin: Unknown | 1
Height [Median (Full Range); unit: cm] | 163 [88 to 186]
Weight [Median (Full Range); unit: kg] | 62 [7.6 to 104]
Body mass index [Median (Full Range); unit: kg/m^2] | 23.5 [13.6 to 40.9]
Family history of Von Willebrand Disease (VWD) [Count of Participants; unit: Participants]
  Yes | 60
  No | 36
  Unknown | 15
Time since diagnosis [Median (Full Range); unit: years] | 5 [0 to 60]
Type of VWD [Count of Participants; unit: Participants] — Von Willebrand disease (VWD) is a genetic bleeding disorder caused by missing or defective von Willebrand factor (VWF) which is a clotting protein. There are three types of VWD: Type 1, 2 and 3. Type 1 VWD patients have a quantitative deficiency of VWF. Levels of VWF in the blood range from 20%-50% of normal; symptoms are usually mild. Type 2 VWD patients have a qualitative deficiency in VWF. Symptoms are mild to moderate. Type 3 VWD patients have a quantitative deficiency of VWF. Symptoms are typically severe, and include spontaneous bleeding episodes, often into their joints and muscles.
  Participants
    Type 1 VWD | 50
    Type 2 VWD | 32
    Type 3 VWD | 20
    Not available | 8
    Not applicable | 1
History of Von Willebrand Factor (VWF) inhibitor activity [Count of Participants; unit: Participants]
  Yes | 1
  No | 83
  Unknown | 27
Known gene mutation [Count of Participants; unit: Participants]
  Yes | 12
  No | 49
  Unknown | 50
Prestudy exposure to Factor VIII (FVIII)/Von Willebrand factor (VWF) products in exposure days (ED)s [Count of Participants; unit: Participants]
  0 | 37
  < 150 EDs | 57
  ≥ 150 EDs | 14
  Not available | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Drug Reactions (ADRs) (%)
Description: Medical Dictionary for Regulatory Activities (MedDRA) primary system organ class preferred term. Incidence rate = number of patients reporting the event / number of patients * 100
Time Frame: Throughout the duration of each patient's participation in the study (mean [± standard deviation (SD)]: 575 days [±326]; median [range]: 731 days [2-1185])
Population: All patients who received at least one dose of Wilate during the study (SAF population).
Measure: Count of Participants; unit: Participants
Groups:
- SAF Population: All patients treated with at least one dose of Wilate during the study.
Arm/Group | SAF Population
Number analyzed (Participants) | 111
Participants
  Any adverse event | 8
  Infections and infestations | 1
  Nervous system disorders | 1
  Cardiac disorders | 3
  Vascular disorders | 2
  Respiratory, thoracic and mediastinal disorders | 2
  Gastrointestinal disorders | 3
  Skin and subcutaneous tissue disorders | 3
  General disorders & administration site conditions | 5

2. Primary Outcome: Tolerability Assessment of Wilate Infusions by Reason for Administration
Description: Tolerability was assessed using a 3-point verbal rating scale (excellent; satisfactory; unsatisfactory) according to overall feeling during and after Wilate therapy and occurrence of ADRs.
  Tolerability was assessed for infusions given for on-demand and prophylactic treatment, but not for infusions administered for surgeries or for the purpose of thrombogenicity assessment. In some instances, however, investigators also recorded the tolerability of infusions given for surgical prophylaxis. For infusions administered for surgeries, only those with available tolerability assessments are presented. Wilate infusion may have been administered to a patient for more than one reason and may be included in more than one category (e.g., if a patient was under Wilate prophylaxis, they could also receive Wilate for the treatment of a bleeding episode [BE] or surgery or menstruation).
Time Frame: During and immediately after each infusion of Wilate during the study.
Population: The tolerability analysis was performed in the SAF population; however, not all of the 111 participants experienced bleeding or had surgery or menstruation.
Measure: Count of Units; unit: Infusions
Units Other Than Participants: Infusions
Groups:
- Prophylaxis: Wilate administered to patients in the context of prophylactic treatment.
- Bleeding: Wilate administered for the treatment of acute or breakthrough BEs (does not include menstrual BEs).
- Surgery: Wilate administered in the context of surgery.
- Menstruation: Wilate administered in the context of menstrual BEs.
- Prevention: Wilate administered for the purpose of preventing recurrent BEs in patients undergoing on-demand treatment or short-term prophylaxis in surgery only.
Arm/Group | Prophylaxis | Bleeding | Surgery | Menstruation | Prevention
Number analyzed (Participants) | 25 | 49 | 62 | 9 | 8
Number analyzed (Infusions) | 5494 | 709 | 44 | 162 | 88
Infusions
  Excellent | 5393 | 654 | 42 | 127 | 38
  Satisfactory | 97 | 55 | 1 | 35 | 50
  Unsatisfactory | 4 | 0 | 1 | 0 | 0

3. Secondary Outcome: Patient and Investigator Efficacy Analysis Assessment of the Treatment of Bleeding Episodes (BEs)
Description: Document the efficacy of Wilate in the treatment of acute BEs, breakthrough BEs in patients receiving prophylactic treatment, and menstrual BEs.
  Efficacy was rated on a 4-point scale (excellent; good; moderate; none) according to overall haemostasis.
Time Frame: During and immediately after treatment of each BE.
Population: From all the patients in the EFF population, 58 patients experienced one or more evaluable BEs; 24 patients experienced acute BEs, 25 patients experienced breakthrough BEs and 9 experienced menstrual BEs.
Measure: Count of Units; unit: Bleeding Episodes (BEs)
Units Other Than Participants: Bleeding Episodes (BEs)
Groups:
- Patient Assessment of Acute BEs: Patient assessment of the efficacy of Wilate in the treatment of acute BEs.
- Investigator Assessment of Acute BEs: Investigator assessment of the efficacy of Wilate in the treatment of acute BEs.
- Patient Assessment of Breakthrough BEs: Patient assessment of the efficacy of Wilate in the treatment of breakthrough BEs.
- Investigator Assessment of Breakthrough BEs: Investigator assessment on the efficacy of Wilate in the treatment of breakthrough BEs.
- Patient Assessment of Menstrual BEs: Patient assessment on the efficacy of Wilate in the treatment of menstrual BEs.
- Investigator Assessment of Menstrual BEs: Investigator assessment on the efficacy of Wilate in the treatment of menstrual BEs.
Arm/Group | Patient Assessment of Acute BEs | Investigator Assessment of Acute BEs | Patient Assessment of Breakthrough BEs | Investigator Assessment of Breakthrough BEs | Patient Assessment of Menstrual BEs | Investigator Assessment of Menstrual BEs
Number analyzed (Participants) | 24 | 24 | 25 | 25 | 9 | 9
Number analyzed (Bleeding Episodes (BEs)) | 136 | 127 | 154 | 139 | 48 | 34
Bleeding Episodes (BEs)
  Excellent | 100 | 94 | 119 | 69 | 23 | 14
  Good | 36 | 33 | 32 | 68 | 17 | 12
  Moderate | 0 | 0 | 3 | 2 | 8 | 8
  None | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Efficacy Analysis for the Prevention of Breakthrough Bleeds During Prophylaxis
Description: Efficacy was rated on a 4-point scale (excellent; good; moderate; none) according to the number of breakthrough bleeds per month. The treatment regimen for prophylactic treatment was at the discretion of the investigator and differed for each patient, as did the duration of prophylactic treatment. The prophylaxis efficacy population (EFF-P) was subdivided into 2 groups, prophylaxis on a continuous basis (EFF-PC population) and prophylaxis on an intermittent basis (EFF-PI population). In total, 25 patients received Wilate for prophylaxis and of these, 17 patients received prophylaxis on a continuous basis, which was defined as: (1) patients having received continuous prophylaxis over a period of at least 3 months, with no treatment gaps longer than 14 days; or (2) patients having received continuous prophylaxis for at least 1 year with an average of 1 infusion/per week (these patients may have had gaps of more than 14 days).
Time Frame: At the end of the study for each patient (study duration: mean [±SD]: 805 days [±247]; median [range]: 797 days [144-1185]).
Population: The efficacy results for the 17 patients with continuous prophylaxis are described here (EFF-PC population).
Measure: Count of Participants; unit: Participants
Groups:
- Spontaneous: Spontaneous bleeding causes
- All Causes: All causes of bleeding episodes
Arm/Group | Spontaneous | All Causes
Number analyzed (Participants) | 17 | 17
Participants
  Excellent (<0.75 breakthrough bleeds per month) | 15 | 12
  Good (0.75-1 breakthrough bleeds per month) | 1 | 2
  Moderate (1-1.5 breakthrough bleeds per month) | 0 | 1
  Poor (>1.5 breakthrough bleeds per month) | 1 | 2

5. Secondary Outcome: Efficacy Analysis of Surgical Prophylaxis
Description: Efficacy was rated on a 4-point scale (excellent; good; moderate; none) according to overall haemostasis during and after surgery.
Time Frame: During and immediately after each surgery.
Population: All patients in the EFF population who underwent surgery under the cover of Wilate (efficacy subpopulation undergoing surgery (EFF-S) population), divided according to surgery type. Efficacy assessments were available for 51/52 minor and 46/46 major surgeries.
Measure: Count of Units; unit: Surgeries
Units Other Than Participants: Surgeries
Groups:
- Minor Surgeries: Efficacy analysis for minor surgeries including treatment with Wilate.
- Major Surgeries: Efficacy analysis for major surgeries including treatment with Wilate.
Arm/Group | Minor Surgeries | Major Surgeries
Number analyzed (Participants) | 62 | 62
Number analyzed (Surgeries) | 51 | 46
Surgeries
  Excellent | 47 | 40
  Good | 3 | 6
  Moderate | 1 | 0
  None | 0 | 0

6. Secondary Outcome: Overall Efficacy Assessment by Patient and Physician at the End of the Treatment Period
Description: Patient and investigator assessment of the overall efficacy of Wilate performed at the end of the study for each patient. Efficacy was rated on a 4-point scale (excellent; good; moderate; none); criteria for assessment were not defined.
Time Frame: At the end of the study for each patient (study duration: mean [±SD]: 596 days [±336]; median [range]: 732 days [2-1185]).
Population: Overall efficacy assessments in the EFF population (n=91) were available from 78 patients, and investigator assessments were available for 86 patients.
Measure: Count of Participants; unit: Participants
Groups:
- Patients: Patient assessment of Wilate efficacy
- Investigator: Investigator assessment of Wilate efficacy
Arm/Group | Patients | Investigator
Number analyzed (Participants) | 78 | 86
Participants
  Excellent | 67 | 71
  Good | 10 | 15
  Moderate | 1 | 0
  None | 0 | 0

7. Other Pre Specified Outcome: Safety: Number of Exposure Days to Wilate
Description: Number of exposure days to Wilate was documented throughout the observation period
  EDs = exposure days. IU = international unit. SD = standard deviation.
Time Frame: Throughout the duration of each patient's participation in the study (study duration: mean [±SD]: 575 days [±326]; median [range]: 731 days [2-1185]).
Population: All patients who received at least one dose of Wilate during the study (SAF Population).
Measure: Median (Full Range); unit: Exposure days
Groups:
- Number of EDs: Number of exposure days
Arm/Group | Number of EDs
Number analyzed (Participants) | 111
Exposure days | 10 [1 to 512]

8. Other Pre Specified Outcome: Safety: Frequency of VWF Inhibitors at Baseline and Follow up
Description: Optional testing for anti-VWF antibodies/VWF inhibitor was performed at the baseline and follow up visits. VWF inhibitor testing was only performed if anti-VWF antibody results were positive. VWF antibody testing was performed using an ELISA assay, and inhibitor testing using a Bethesda assay. Both assays were considered experimental, since no standardized laboratory assays were available. Results displayed here are for confirmatory inhibitor testing.
Time Frame: Optional antibody tests were performed at baseline and 3-4 days (preferable 7 days) after Wilate injection.
Population: Data was analysed for all patients in the SAF population who underwent VWF inhibitor testing. Results were not available at all visits for all patients.
Measure: Count of Participants; unit: Participants
Groups:
- Baseline: Inhibitor results from patients at baseline
- Follow-up: Inhibitor results from patients at follow-up
Arm/Group | Baseline | Follow-up
Number analyzed (Participants) | 17 | 20
Participants
  Positive confirmatory inhibitor results | 1 | 4
  Negative confirmatory inhibitor results | 15 | 16
  Confirmatory inhibitor results not done | 1 | 0

9. Other Pre Specified Outcome: Adverse Drug Reactions (ADRs)
Description: Patients with a positive inhibitor test were assessed for ADRs related to anti VWF antibody or inhibitor development
Time Frame: Optional antibody tests were performed at baseline and 3-4 days (preferable 7 days) after Wilate injection
Population: ADRs were assessed for all patients who has a positive VWF inhibitor testing result as described in outcome 8.
Measure: Number; unit: Adverse drug reactions
Arm/Group | Baseline | Follow-up
Number analyzed (Participants) | 1 | 4
Adverse drug reactions | 0 | 0

10. Other Pre Specified Outcome: Safety: Patients With Thrombogenicity Values >2 Times the Upper Limit of Normal (ULN)
Description: Thrombogenicity testing was optional. Thrombogenicity markers (prothrombin fragments 1 + 2; D-dimer) were evaluated at baseline and during follow up. Samples with prothrombin F1+2 and/or D-dimer values at least 2 times above the upper limit of normal were recorded as high.
Time Frame: Optional thrombogenicity tests were performed at baseline and 1, 3 and 24 hours after each administration of Wilate.
Population: A total of 47 patients were assessed over multiple visits. Results were not available at all visits for all patients.
Measure: Count of Participants; unit: Participants
Groups:
- Prothrombin (Pre-infusion): Pre-infusion assessment of prothrombin F1 + 2 (>2-fold ULN)
- Prothrombin (Post-infusion): Post-infusion assessment of prothrombin F1 + 2 (>2-fold ULN)
- D-Dimer (Pre-infusion): Pre-infusion assessment of D-dimer (>2-fold ULN)
- D-Dimer (Post-infusion): Post-infusion assessment of D-dimer (>2-fold ULN)
Arm/Group | Prothrombin (Pre-infusion) | Prothrombin (Post-infusion) | D-Dimer (Pre-infusion) | D-Dimer (Post-infusion)
Number analyzed (Participants) | 46 | 46 | 46 | 46
Participants
  Number of patients | 10 | 17 | 3 | 6
  No sample available | 1 | 0 | 0 | 0

11. Other Pre Specified Outcome: Wilate Dosage Per Infusion for the Treatment of Acute Bleeding Episodes (BEs; On-demand)
Description: The number of infusions and dosage of Wilate administered for the on-demand treatment of acute BEs was documented throughout the study.
  n= number of infusions
Time Frame: Throughout the duration of each patient's participation in the study (study duration: mean [±SD]: 677 days [±264]; median [range]: 749 days [40-1052]).
Population: Bleeding episodes (BEs) occurring in the efficacy on-demand (EFF-OD) population that included 25 patients. Menstrual BEs were excluded from this analysis.
Measure: Median (Full Range); unit: IU/kg per infusion
Units Other Than Participants: Number of infusions
Groups:
- Dose of Wilate Per Infusion, IU/kg Per Infusion: Dose of Wilate given on-demand per infusion, units per kg per infusion
Arm/Group | Dose of Wilate Per Infusion, IU/kg Per Infusion
Number analyzed (Participants) | 25
Number analyzed (Number of infusions) | 206
IU/kg per infusion | 31.7 [5.6 to 87.7]

12. Other Pre Specified Outcome: Wilate Dosage for the Treatment of Acute Bleeding Episodes (BEs; On-demand) Per Bleeding Episode (BE)
Description: The dosage of Wilate administered for the on-demand treatment of acute BEs was documented throughout the study.
  n = number of BEs
Time Frame: as for outcome 11
Population: Bleeding episodes (BEs) occurring in the efficacy on-demand (EFF-OD) population that included 25 patients.
Measure: Median (Full Range); unit: IU/kg per BE
Units Other Than Participants: Number of BEs
Groups:
- Dose of Wilate Per BE, IU/kg Per BE: Dose of Wilate given on-demand per BE
Arm/Group | Dose of Wilate Per BE, IU/kg Per BE
Number analyzed (Participants) | 25
Number analyzed (Number of BEs) | 136
IU/kg per BE | 33 [8.2 to 625]

13. Other Pre Specified Outcome: Wilate Doses for the Treatment of Menstrual Bleeding Episodes (BEs)
Description: Dosage of Wilate administered for treatment of menstrual BE's was documented throughout the study.
  n = number of BEs treated
Time Frame: Throughout the duration of each patient's participation in the study (study duration: mean [±SD]: 553 days [±296]; median [range]: 713 days [125-840]).
Population: Nine patients from the EFF population had a total of 56 menstrual BEs treated with Wilate.
Measure: Median (Full Range); unit: IU/kg per menstrual BE
Units Other Than Participants: Number of menstrual BEs
Groups:
- Dose of Wilate Per Menstrual BE, IU/kg Per Menstrual BE: Dose of Wilate given to participants per menstrual BE, units per kg per menstrual BE
Arm/Group | Dose of Wilate Per Menstrual BE, IU/kg Per Menstrual BE
Number analyzed (Participants) | 9
Number analyzed (Number of menstrual BEs) | 56
IU/kg per menstrual BE | 79.1 [10 to 339.8]

14. Other Pre Specified Outcome: Exposure Days for Prophylactic Treatment With Wilate
Description: The treatment regimen for prophylactic treatment was at the discretion of the investigator and differed for each patient, as did the duration of prophylactic treatment. The prophylaxis efficacy population (EFF-P) was subdivided into 2 groups, prophylaxis on a continuous basis (EFF-PC population) and prophylaxis on an intermittent basis (EFF-PI population).
Time Frame: Throughout the duration of each patient's participation in the study (study duration: mean [±SD]: 761 days [±251]; median [range]: 773 days [144-1185]).
Population: Patients receiving prophylactic treatment (n=25) on either a continuous basis (EFF-PC population) or an intermittent basis (EFF-PI population).
Measure: Median (Full Range); unit: Exposure days
Groups:
- Number of Exposure Days: Number of prophylactic exposure days.
Arm/Group | Number of Exposure Days
Number analyzed (Participants) | 25
Exposure days | 145 [11 to 512]

15. Other Pre Specified Outcome: Number of Infusions of Prophylactic Treatment With Wilate Per Week
Description: The treatment regimen for prophylactic treatment was at the discretion of the investigator and differed for each patient, as did the duration of prophylactic treatment. The prophylaxis efficacy population (EFF-P) was subdivided into 2 groups, prophylaxis on a continuous basis (EFF-PC population) and prophylaxis on an intermittent basis (EFF-PI population).
  n = number of patients.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: Infusions per week
Groups:
- Number of Wilate Infusions Per Week: The number of prophylactic Wilate infusions given to participants per week.
Arm/Group | Number of Wilate Infusions Per Week
Number analyzed (Participants) | 25
Infusions per week | 2 [0.5 to 4.2]

16. Other Pre Specified Outcome: Dosage for Prophylactic Treatment With Wilate Per Week
Description: as for outcome 15
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: IU/kg per week
Groups:
- Dose of Wilate Per Week, IU/kg Per Week: The prophylactic dose of Wilate given to participants per week
Arm/Group | Dose of Wilate Per Week, IU/kg Per Week
Number analyzed (Participants) | 25
IU/kg per week | 69.3 [8.2 to 298.6]

17. Other Pre Specified Outcome: Dosage for Prophylactic Treatment With Wilate Per Infusion
Description: as for outcome 14
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: IU/kg per infusion
Units Other Than Participants: Number of infusions
Groups:
- Dose of Wilate Per Infusion, IU/kg Per Infusion: Dose of prophylactic Wilate administered per infusion
Arm/Group | Dose of Wilate Per Infusion, IU/kg Per Infusion
Number analyzed (Participants) | 25
Number analyzed (Number of infusions) | 4584
IU/kg per infusion | 31.3 [8.3 to 183.7]

18. Other Pre Specified Outcome: Exposure Days for Prophylactic Wilate Treatment on a Continuous Basis
Description: Number and dosage of Wilate infusions administered as prophylactic treatment on a continuous basis were documented throughout the study.
  The treatment regimen for prophylactic treatment was at the discretion of the investigator and differed for each patient, as did the duration of prophylactic treatment.
Time Frame: Throughout the duration of each patient's participation in the study (study duration: mean [±SD]: 805 days [±247]; median [range]: 797 days [144-1185]).
Population: Patients receiving prophylactic Wilate (n=17) on a continuous basis (EFF-PC population).
Measure: Median (Full Range); unit: Exposure days
Groups:
- Number of Exposure Days (EDs): Number of prophylactic exposure days
Arm/Group | Number of Exposure Days (EDs)
Number analyzed (Participants) | 17
Exposure days | 271 [36 to 512]

19. Other Pre Specified Outcome: Number of Infusions Per Week for Prophylactic Wilate Treatment on a Continuous Basis
Description: as for outcome 18
Time Frame: as for outcome 18
Population: Patients receiving prophylactic Wilate (n=17) on a continuous basis (EFF-PC population).
Measure: Median (Full Range); unit: Infusions per week
Groups:
- Number of Wilate Infusions Per Week: The prophylactic dose of Wilate given to participants per week
Arm/Group | Number of Wilate Infusions Per Week
Number analyzed (Participants) | 17
Infusions per week | 2.6 [1 to 4.2]

20. Other Pre Specified Outcome: Dosage for Prophylactic Wilate Treatment on a Continuous Basis
Description: Number and dosage of Wilate infusions administered as prophylactic treatment on a continuous basis were documented throughout the study.
  The treatment regimen for prophylactic treatment was at the discretion of the investigator and differed for each patient, as did the duration of prophylactic treatment.
  n = number of patients.
Time Frame: as for outcome 18
Population: Patients receiving prophylactic Wilate (n=17) on a continuous basis (EFF-PC population).
Measure: Median (Full Range); unit: IU/kg per week
Groups:
- Dose of Wilate Per Week, IU/kg Per Week: The prophylactic dose of Wilate given to participants per week, per kg
Arm/Group | Dose of Wilate Per Week, IU/kg Per Week
Number analyzed (Participants) | 17
IU/kg per week | 77.5 [19.3 to 201.3]

21. Other Pre Specified Outcome: Dosage for Prophylactic Wilate Treatment Per Infusion on a Continuous Basis
Description: Number and dosage of Wilate infusions administered as prophylactic treatment on a continuous basis were documented throughout the study.
  The treatment regimen for prophylactic treatment was at the discretion of the investigator and differed for each patient, as did the duration of prophylactic treatment.
  n = number of infusions.
Time Frame: as for outcome 18
Population: Patients receiving prophylactic Wilate (n=17) on a continuous basis (EFF-PC population).
Measure: Median (Full Range); unit: IU/kg per infusion
Units Other Than Participants: Number of infusions
Groups:
- Dose of Wilate Per Infusion, IU/kg Per Infusion: The prophylactic dose of Wilate given to participants per infusion, per kg per infusion
Arm/Group | Dose of Wilate Per Infusion, IU/kg Per Infusion
Number analyzed (Participants) | 17
Number analyzed (Number of infusions) | 4120
IU/kg per infusion | 31.3 [8.3 to 111.1]

22. Other Pre Specified Outcome: Dosage of Wilate Per Infusion for the Treatment of Breakthrough Bleeds
Description: Number and dosage of Wilate infusions administered as treatment for breakthrough bleeds in patients receiving prophylactic treatment on a continuous or intermittent basis were documented throughout the study. n = number of infusions
Time Frame: Throughout the duration of each patient's participation in the study (study duration: mean [±SD]: 561 days [±251]; median [range]: 773 days [144-1185]).
Population: The EFF-P population included 25 patients.
Measure: Median (Full Range); unit: IU/kg per infusion
Units Other Than Participants: Number of infusions
Groups:
- Dose of Wilate Per Infusion, IU/kg Per Infusion: The dose of Wilate given to participants per infusions, per kg to treat breakthrough bleeds
Arm/Group | Dose of Wilate Per Infusion, IU/kg Per Infusion
Number analyzed (Participants) | 25
Number analyzed (Number of infusions) | 292
IU/kg per infusion | 52.4 [8.3 to 125]

23. Other Pre Specified Outcome: Dosage of Wilate for the Treatment of Breakthrough Bleeds Per Breakthrough Bleed
Description: Number and dosage of Wilate infusions administered as treatment for breakthrough bleeds in patients receiving prophylactic treatment on a continuous or intermittent basis were documented throughout the study.
  n = For 1 bleed in the EFF-PC population, the dose is unknown.
Time Frame: as for outcome 22
Population: Treatment of breakthrough bleeds (n=175) in the EFF-P population that included 25 patients.
Measure: Median (Full Range); unit: IU/kg per breakthrough bleed
Units Other Than Participants: No. of breakthrough bleeds
Groups:
- Dose of Wilate Per Breakthrough Bleed: The dose of Wilate given to participants per breakthrough bleed, units per kg per breakthrough bleed
Arm/Group | Dose of Wilate Per Breakthrough Bleed
Number analyzed (Participants) | 25
Number analyzed (No. of breakthrough bleeds) | 175
IU/kg per breakthrough bleed | 55.4 [8.3 to 1441.3]

24. Other Pre Specified Outcome: Wilate Dosage Per Infusion for the Prevention of Bleeding During and After Surgery
Description: Number and dosage of Wilate infusions administered to prevent bleeding during and after surgery were documented throughout the study.
  1. For 6 infusions, no dosage information is available
  2. One minor surgical procedure was not treated with Wilate. For 2 of the 98 treated surgical procedures, no dosage information is available (i.e., 1 major orthopaedic surgery and 1 minor cardiovascular surgery)
Time Frame: Throughout the duration of each patient's participation in the study (study duration: mean [±SD]: 568 days [±349]; median [range]: 732 days [2-1185]).
Population: Efficacy of Wilate for the prevention of bleeding during and after surgery was assessed in the efficacy surgery (EFF-S) population that included 62 patients.
Measure: Median (Full Range); unit: IU/kg per infusion
Units Other Than Participants: Number of infusions
Groups:
- Dose of Wilate Per Infusion, IU/kg Per Infusion: Dose of Wilate per infusion, units per kg in patients following surgery.
Arm/Group | Dose of Wilate Per Infusion, IU/kg Per Infusion
Number analyzed (Participants) | 62
Number analyzed (Number of infusions) | 384
IU/kg per infusion | 27.8 [1.1 to 92.3]

25. Other Pre Specified Outcome: Wilate Dosage Per Procedure for the Prevention of Bleeding During and After Surgery
Description: Number and dosage of Wilate infusions administered to prevent bleeding during and after surgery were documented throughout the study.
  1. For 6 infusions, no dosage information is available
  2. One minor surgical procedure was not treated with Wilate. For 2 of the 98 treated surgical procedures, no dosage information is available (i.e., 1 major orthopedic surgery and 1 minor cardiovascular surgery)
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Median (Full Range); unit: IU/kg per procedure
Units Other Than Participants: Number of treated surgeries
Groups:
- Dose of Wilate Per Procedure, IU/kg Per Procedure: Dose of Wilate per procedure, units per kg in patients following surgery
Arm/Group | Dose of Wilate Per Procedure, IU/kg Per Procedure
Number analyzed (Participants) | 62
Number analyzed (Number of treated surgeries) | 96
IU/kg per procedure | 69.2 [6.3 to 679.6]

26. Other Pre Specified Outcome: Number of Patients With Breakthrough Bleeds During Prophylaxis
Description: Breakthrough bleeds in patients receiving Wilate as prophylactic treatment on a continuous (EFF-PC population) or intermittent (EFF-PI population) basis were documented throughout the study.
Time Frame: as for outcome 14
Population: Patients who received Wilate as prophylaxis were sub-divided into those who received prophylaxis on a continuous basis (EFF-PC Population) and those who received prophylaxis on an intermittent basis (EFF-PI).
Measure: Count of Participants; unit: Participants
Groups:
- EFF-PC: Efficacy population undergoing continuous prophylaxis.
- EFF-PI: Efficacy population undergoing intermittent prophylaxis.
Arm/Group | EFF-PC | EFF-PI
Number analyzed (Participants) | 17 | 8
Participants | 13 | 5

27. Post Hoc Outcome: Thromboembolic Adverse Drug Reactions (ADRs)
Description: Patients with elevated F1 + F2 and/or D-dimer levels were monitored for thromboembolic ADRs
Time Frame: Optional thrombogenicity tests were performed at baseline and 1,3 and 24 hours after each administration of Wilate
Population: Thromboembolic ADRs were analysed for all patients who has elevated F1 + F2 and/or D-dimer levels >2 times the upper limit of normal as identified in outcome 11.
Measure: Number; unit: number of adverse drug reactions
Arm/Group | Prothrombin (Pre-infusion) | Prothrombin (Post-infusion) | D-Dimer (Pre-infusion) | D-Dimer (Post-infusion)
Number analyzed (Participants) | 10 | 17 | 3 | 6
number of adverse drug reactions | 0 | 0 | 0 | 0

28. Post Hoc Outcome: Clinical Symptoms of Von Willebrand Factor (VWF) Inhibition
Description: Patients with a positive inhibitor tests were assessed for clinical symptoms of VWF inhibition
Time Frame: Optional antibody tests were performed at baseline and 3-4 days (preferable 7 days) after Wilate injection
Population: Data was assessed for all patients in the SAF population who had a positive VWF inhibitor testing result as described in outcome 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | Follow-up
Number analyzed (Participants) | 1 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the duration of each patient's participation in the study (study duration: mean [±SD]: 575 days [±326]; median [range]: 731 days [2-1185]).
Groups:
- SAF Population: All patients who received at least one dose of Wilate during the study.
Arm/Group | SAF Population
All-Cause Mortality (participants affected / at risk) | 0/111
Serious Adverse Events (participants affected / at risk) | 0/111
Other Adverse Events (participants affected / at risk) | 8/111
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAF Population (N=111)
Erythema Infectiosum (Infections and infestations) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3)
Flushing (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Administration Site Reaction (General disorders) | 1 (1)
Chest Discomfort (General disorders) | 1 (1)
Drug Ineffective (General disorders) | 1 (1)
Face Oedema (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Injection Site Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-08-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT01602419/Prot_002.pdf
  • Statistical Analysis Plan (2015-12-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT01602419/SAP_003.pdf